CLINICAL TRIAL: NCT00437112
Title: A Phase 3, Open-Label, Crossover Study to Evaluate the Efficacy and Safety of Human Insulin Inhalation Powder (HIIP) Compared With Once-Daily Insulin Glargine in Insulin-Naive Patients With Type 2 Diabetes Mellitus on Oral Agents
Brief Title: Evaluate the Efficacy and Safety of Insulin Compared to Glargine in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9631; H7U-MC-IDAZ
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (2):
- 1 (Experimental): 4 week pretreatment phase consists of continuation of usual OAM therapy
  24 week treatment period with insulin glargine and OAM continuation followed by 24 week treatment period with HIIP and OAM continuation
  8 week follow up period
  Interventions: Drug: Human Insulin Inhalation Powder; Drug: Insulin Glargine
- 2 (Experimental): 4 week pretreatment phase consists of continuation of usual OAM therapy
  24 week treatment period with HIIP and OAM continuation followed by 24 week treatment period with insulin glargine and OAM continuation
  8 week follow up period
  Interventions: Drug: Human Insulin Inhalation Powder; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Human Insulin Inhalation Powder — patient specific dose, inhaled, before meals, 24 weeks
  Other Names: LY041001
Drug: Insulin Glargine — patient specific dose, injectable, before meals, 24 weeks

SUMMARY:
A study to compare Human Inhalation Powder (also known as AIR® Inhaled Insulin) (AIR® is a registered trademark of Alkermes, Inc.)with insulin glargine injections in patients with Type 2 diabetes who are currently taking oral medications and have not previously taken insulin. Change in HbA1c levels will be reviewed to determine superiority or inferiority of the AIR Inhaled Insulin regimen.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Insulin naive
* One or more oral antihyperglycemic medications
* HbA1c greater than or equal to 8.0% and less than or equal to 10.5%
* Non-smoker

Exclusion Criteria:

* Taking a TZD dose greater than what is indicated
* Have not taken insulin within 6 months of entry into study
* Have had more than 2 episodes of sever hypoglycemia during the 6 months prior to study entry
* Have had more than 1 hospitalization or emergency room visit due to poor diabetic control during the 6 months prior to study entry
* Have had pneumonia in the 3 months prior to study entry
* Systemic glucocorticoid therapy
* Clinical signs or symptoms of liver disease, acute or chronic hepatitis
* History of renal transplantation
* Have an active or untreated malignancy
* Have a current diagnosis or past history of clinically relevant pulmonary disease
* Taking or have taken exenatide during the 6 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Compare, in insulin-naive patients with type 2 diabetes on one or more oral antihyperglycemic medications, a regimen adding mealtime HIIP versus a regimen adding insulin glargine with respect to change in HbA1c from baseline to endpoint. | 56 weeks

SECONDARY OUTCOMES:
Mean change in HbA1c from baseline to various timepoints | 56 weeks
Insulin dose requirements | 56 weeks
Patient-reported outcomes of W-BQ12 | screening,baseline, week 12,24, and 48
Hypoglycemia rate | throughout the study
Changes in body weight | every visit
Adverse events | throughout the study
Safety as assessed by total pulmonary function testing and fasting lipid profile | throughout the study
Assess inhaler reliability. | throughout the study
Patient Reported outcomes of DSC-R | screening,baseline, week 12,24, and 48
Patient reported outcomes of DTSQS | screening,baseline, week 12, 24 and 48
Patient reported outcome of IDSQ | week 12, 24, and 48
Patient reported outcome of preference questionnaire | week 48
Patient reported outcome of Expectations About Insulin Therapy Questionnaire | screening,baseline
Patient reported outcome of Experience with Insulin Therapy Questionnaire | week 12, 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri from 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Braunfels, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vellore
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barakaldo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dos Hermanas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Requena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell

REFERENCES:
- See also: Lilly CSR Synopsis — https://www.lilly.com/clinical-study-report-csr-synopses